CLINICAL TRIAL: NCT02509637
Title: Acute Effects of a Flutter Device and Chest Wall Compression on Respiratory System Impedance in Bronchiectasis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Ada Clarice Gastaldi, PhD, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: USP 2015-3
Record Dates: First submitted 2015-07-03; First posted 2015-07-28 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Bronchiectasis
Keywords: Respiratory System; Physical Therapy Modalities
MeSH Terms: conditions — Bronchiectasis | interventions — Chest Wall Oscillation; Drug Tolerance; Oximetry

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Flutter Intervention (Active Comparator): After initial evaluation, the subjects will perform breathing exercises with quiet inspiration and prolonged expiration on the device for thirty minutes, with breaks of one minute every four minutes. Immediately after the exercise will be performed new assessment against Impulse Oscillometry. Then patients will be kept for 30 minutes at rest and at the end will be applied the acceptability and tolerance scale and a third evaluation with Impulse Oscillometry. The secretions expectorated during the protocol will be evaluated for weight, adhesiveness and purulence.
  Interventions: Device: Flutter; Other: Impulse Oscillometric; Other: Dyspnea scale; Other: Acceptability and tolerance; Device: Pulse oximetry; Other: Difficulty sputum
- Chest Compression Intervention (Active Comparator): After initial evaluation, the subjects will be instructed to perform deep breaths between three quiet inspiration brought, and expiration will be accompanied by bilateral compression with the therapist's hands on the lower ribs during thirty minutes with one minute intervals of rest every four minutes. Immediately after the exercise will be performed new assessment against Impulse Oscillometry. Then patients will be kept for 30 minutes at rest and at the end will be applied the acceptability and tolerance scale and a third evaluation with Impulse Oscillometry. The secretions expectorated during the protocol will be evaluated for weight, adhesiveness and purulence.
  Interventions: Other: Chest Compression; Other: Impulse Oscillometric; Other: Dyspnea scale; Other: Acceptability and tolerance; Device: Pulse oximetry; Other: Difficulty sputum
- Crontrol Intervention (Active Comparator): After initial evaluation, patients will be remain seated quiet breathing without any guidance for thirty minutes. Immediately after this time will be held reassessment with Impulse Oscillometry. Then patients will be kept for 30 minutes at rest and at the end will be applied to acceptance and tolerance scale and a third evaluation with Impulse Oscillometry. The secretions expectorated during the protocol will be evaluated for wight, adhesiveness and purulence.
  Interventions: Other: Control; Other: Impulse Oscillometric; Other: Dyspnea scale; Other: Acceptability and tolerance; Device: Pulse oximetry; Other: Difficulty sputum

INTERVENTIONS:
Device: Flutter — Flutter is a small device, simple, like a plastic pipe with a mouthpiece at one end and a perforated cover on the other, containing a steel ball resting in a plastic cone inside. When the patient exhales through the flutter expiratory flow causes movement of the ball, creating an oscillatory positive pressure.
  Arms: Flutter Intervention
Other: Chest Compression — Manual chest compression is based on the application of forces resulting from the action of respiratory muscles or physiotherapist manual action in order to increase the alveolar pressure creating a pressure gradient to promote change in pulmonary flow and volume.It consists of vigorous compression of the chest at the beginning of expiration or during expiration.
  Arms: Chest Compression Intervention
Other: Control
  Arms: Crontrol Intervention
Other: Impulse Oscillometric — For this measure will be used IOS Jaeger (Jaeger, Wurzburg, Germany). to minimize the effect of the bad positioning of the tongue will use a mouth "free-flow", which contains a depressant for keeping the tongue in the mouth soil, stabilizing it and reducing oral resistance. Volunteers will support hands firmly on the cheeks to reduce the effect of oscillation thereof. The measures will be carried out with the volunteer sitting, using nasal, relaxed and your head in neutral clip, breathing normally through the mouthpiece to his lips tightly sealed to prevent air leaks.
Other: Dyspnea scale — Dyspnea will be evaluated across the range Medical Research Council (MRC) for use in patients with chronic obstructive pulmonary disease in Brazil.
Other: Acceptability and tolerance — patients will complete scales 1-7, 1: extremely and 7: none) on usefulness, ease to understand the instructions, easy to perform the exercises, degree of fatigue and discomfort
Device: Pulse oximetry — During therapy the patient will remain monitored with digital oximeter and the information will be recorded before and after the procedures
Other: Difficulty sputum — Patients inform the ease or difficulty sputum according to a scale of 1 to 5, where 1 = no difficulty and 5 = extremely difficult.

SUMMARY:
Bronchiectasis is characterized pathologically by the abnormal and permanent dilation of bronchi caused mainly by the perpetuation of inflammation and impaired clearance of secretions. Physical therapy is essential in the treatment of these patients, using its various techniques and devices. The aim of this study is to evaluate the impedance of the respiratory system, by impulse oscillometry, after breathing exercises with chest compression or flutter in patients with bronchiectasis, considering that there are no results in the literature on the effect of these techniques in the small airways of these patients.

DETAILED DESCRIPTION:
Bronchiectasis patients and healthy subjects will be evaluated before and after a 30 minutes session of control, breathing exercises with flutter valve, that is a device that produces oscillation and positive pressure during the expiratory phase, or chest compression, that is a manual manoeuvre in the right and left sides of the lower chest, all of them in a sitting position. The main outcome will be obtained by impulse oscillometry, that is a method to access large and small airways, to evaluate the resistance (R), reactance (X), reactance area (AX) and resonant frequency (Fres) of respiratory system for the whole breath and for inspiratory and expiratory phase. Additionally, will be analysed the dyspnea using the Medical Research Council scale; acceptability and tolerability scale; pulse oxymetry; difficulty of expectoration score; and volume, adhesivity and purulence of sputum.

ELIGIBILITY:
Inclusion Criteria:

* aged between 30 and 80 years
* diagnosed with bronchiectasis not resulting from cystic fibrosis, defined by history and full clinical examination and confirmed by computed tomography.

Exclusion Criteria:

* Chest pain
* acute hemoptysis
* recent history rib fracture and pneumothorax
* respiratory infection in the last 4 weeks prior to study
* cystic fibrosis
* asthma
* fistula.
* chronic obstructive pulmonary disease

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Respiratory System Impedance | In the primary evaluation, and after seven and fourteen days.
  Will be evaluated the resistance (R), reactance (X), reactance area (AX) and resonance frequency (Fres) before, immediately after the intervention and after 30 minutes of rest in order of identifying changes in the components of resistance of airways of individuals.
Difficulty sputum | In the primary evaluation, and after seven and fourteen days.
  Patients inform the ease or difficulty in expectoration in accordance with a scale of 1 to 5, where 1 = no difficulty and 5 = extremely difficult. (Burioka, 1998). The scale will be applied at baseline and always after the intervention to assess whether there is difference in the difficulty of sputum between sessions.
Secretions weight | In the primary evaluation, and after seven and fourteen days.
  The secretions are collected in the universal and heavy collectors on a precision balance.They will be evaluated in the total weight measurements and a dry weight and wet mucus. The weight of mucus of each interventions are compared to determine a technique with improved efficiency for removal of secretions.

SECONDARY OUTCOMES:
Pulse oximetry | In the primary evaluation, and after seven and fourteen days.
  During therapy the patient will remain monitored with digital oximeter and the information will be recorded before and after the procedures
Acceptability and tolerance | In the primary evaluation, and after seven and fourteen days.
  30 minutes after the treatment session or control, patients will complete scales 1-7, 1: extremely and 7: none) on usefulness, ease to understand the instructions, easy to perform the exercises, degree of fatigue and discomfort (adapted EATON, 2007).
Dyspnea scale: | In the primary evaluation, and after seven and fourteen days.
  Dyspnea will be evaluated across the range Medical Research Council (MRC) for use in patients with chronic obstructive pulmonary disease in Brazil. The MRC scale comprises only five items, and the patient chooses the item corresponding to as dyspnea limits their activities of daily living. The patient reports its subjective degree of dyspnea choosing a value ranging from 1 to 5, with 1 (only suffers from shortness of breath during intense exercise), 2 (suffers from shortness of breath when walking briskly or climbing a slight slope) 3 (walks slower than people of the same age because of breathlessness or has to stop for breath even when walking slowly), 4 (stops for breath after walking less than 100 m or after a few minutes) and 5 (feel so short of breath that does not go over the house, or feel short of breath when getting dressed) (KOLEVIS et al., 2008).
Adhesiveness of expectorated secretion: | In the primary evaluation, and after seven and fourteen days.
  Immediately after the separation of secretion with saliva, mucus will be evaluated for its adhesion award a note according to visual scale described by Lopez-Vidriero et al., 1973. Test samples giving the adhesive index between 1 (fully adhered) and 2 (small movement under gravity) will be classified as adhesive and between 3 (slow moving mass) and 4 (easy handling) will be classified as non-adhesive.

CONTACTS AND LOCATIONS:
Overall Officials: Ada C Gastaldi, PhD, Principal Investigator — Ribeirão Preto Medicine School - University of São Paulo
Locations (1):
- Ribeirão Preto Medicine School, University of São Paulo, Ribeirão Preto, São Paulo, Brazil

REFERENCES:
- [Background] Tambascio J, de Souza LT, Lisboa RM, Passarelli Rde C, de Souza HC, Gastaldi AC. The influence of Flutter(R)VRP1 components on mucus transport of patients with bronchiectasis. Respir Med. 2011 Sep;105(9):1316-21. doi: 10.1016/j.rmed.2011.04.017. PMID 21641196
- [Background] Oostveen E, MacLeod D, Lorino H, Farre R, Hantos Z, Desager K, Marchal F; ERS Task Force on Respiratory Impedance Measurements. The forced oscillation technique in clinical practice: methodology, recommendations and future developments. Eur Respir J. 2003 Dec;22(6):1026-41. doi: 10.1183/09031936.03.00089403. PMID 14680096
- [Background] Murray MP, Pentland JL, Turnbull K, MacQuarrie S, Hill AT. Sputum colour: a useful clinical tool in non-cystic fibrosis bronchiectasis. Eur Respir J. 2009 Aug;34(2):361-4. doi: 10.1183/09031936.00163208. PMID 19648517
- [Background] McCarren B, Alison JA, Herbert RD. Manual vibration increases expiratory flow rate via increased intrapleural pressure in healthy adults: an experimental study. Aust J Physiother. 2006;52(4):267-71. doi: 10.1016/s0004-9514(06)70006-x. PMID 17132121
- [Result] Eaton T, Young P, Zeng I, Kolbe J. A randomized evaluation of the acute efficacy, acceptability and tolerability of flutter and active cycle of breathing with and without postural drainage in non-cystic fibrosis bronchiectasis. Chron Respir Dis. 2007;4(1):23-30. doi: 10.1177/1479972306074481. PMID 17416150
- [Derived] de Souza Simoni LH, Dos Santos DO, de Souza HCD, Baddini-Martinez JA, Santos MK, Gastaldi AC. Acute Effects of Oscillatory PEP and Thoracic Compression on Secretion Removal and Impedance of the Respiratory System in Non-Cystic Fibrosis Bronchiectasis. Respir Care. 2019 Jul;64(7):818-827. doi: 10.4187/respcare.06025. Epub 2019 May 28. PMID 31138732